CLINICAL TRIAL: NCT06300177
Title: A Randomized, Controlled, Double-blind, Double-simulated, Multicenter Phase III Clinical Study Evaluating D-1553 Tablet Versus Docetaxel Injection for KRAS G12C Mutation-positive Locally Advanced or Metastatic Non-small Cell Lung Cancer After Prior Standard Therapy Failure.
Brief Title: D-1553 Tablet Versus Docetaxel Injection for KRAS G12C Mutation-positive Locally Advanced or Metastatic Non-small Cell Lung Cancer After Prior Standard Therapy Failure
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1553-III-01
Record Dates: First submitted 2024-03-03; First posted 2024-03-08 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-03

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D-1553 Tablet (Experimental): D-1553 Tablet，21 days as a treatment cycle.
  Interventions: Drug: D-1553 Tablet
- Docetaxel Injection (Active Comparator): Docetaxel Injection，21 days as a treatment cycle.
  Interventions: Drug: Docetaxel injection

INTERVENTIONS:
Drug: D-1553 Tablet — D-1553 is a KRAS inhibitor.
  Arms: D-1553 Tablet
Drug: Docetaxel injection — Docetaxel, is an anti-tumor drug, significantly reduces the number of free tubules by promoting tubule polymerization into stable microtubules and inhibiting their depolymerization.
  Arms: Docetaxel Injection

SUMMARY:
The purpose of this project is to evaluate progression-free survival (PFS) of D-1553 Tablet versus Docetaxel Injection in subjects with prior standard therapy failure kirsten rat sarcoma viral oncogene (KRAS) G12C mutation positive locally advanced or metastatic non small cell lung cancer (NSCLC), progression-free survival (PFS) as assessed by the Independent Review Committee (IRC) based on RECIST 1.1 was used as the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in the study and sign of written informed consent after full informed consent, willing and able to comply with the study procedures and requirements specified in the protocol;
* Age greater than or equal to 18 years old; male and female; eastern cooperative oncology group performance status (ECOG) score 0-1; expected survival period greater than or equal to 3 months;
* Pathologically confirmed locally advanced, unresectable and / or metastatic non-small cell lung cancer (stage III b / III c / IV of american joint committee on cancer (AJCC) 8th);
* Subjects must provide adequate and qualified tumor tissue specimens (surgical resection samples or puncture / biopsy tissue samples within 2 years prior to screening) for confirmation of the KRAS G12C mutation in the central laboratory;
* Disease progression or toxicity after previous treatment with first-line anti-PD-1 / PD-L1 and platinum-containing chemotherapy is not tolerated.Subjects who have clear medical reasons and can not tolerate anti-PD-1 / PD-L1 therapy or platinum-containing chemotherapy;
* Having at least one target lesion according to RECIST 1.1;
* Good function of the major organs;
* Female subjects of childbearing age should agree that contraception must be used during the study and within 6 months after the end of the study; the serum pregnancy test is negative within 7 days before study enrollment and must be non-lactating subjects; male subjects should agree that contraception must be used during the study and within 6 months after the end of the study period.

Exclusion Criteria:

* Treatment with a KRAS G12C mutation inhibitor or docetaxel at any previous time;
* NSCLC with mutations of other driver genes;
* Symptomatic or progressive aggravation of central nervous system metastasis or cancerous meningitis. Subjects with a history of brain metastasis may be considered to be selected if they are clinically stable;
* Patients with a previous history of epilepsy；presence of superior vena cava syndrome;
* Cardiovascular system meets any condition:

  1. New York Heart Association (NYHA) Heart Function Grade II and above congestive heart failure;
  2. Severe cardiac arrhythmias requiring medical treatment;
  3. Acute myocardial infarction, severe or unstable angina pectoris, coronary or peripheral artery bypass surgery within 6 months prior to enrollment;
  4. Left ventricular ejection fraction (LVEF) <50%;
  5. QT interval (QTcF) at prolonged;
  6. Hypertension that is not effectively controlled;
* Subjects with stroke or other severe cerebrovascular disease within 6 months before enrollment;
* History of deep vein thrombosis or any other serious thromboembolism within 3 months prior to enrollment;
* History of interstitial lung disease, radiation pneumonitis, and immune-associated pneumonia previously treated with steroids, Or active non-infectious pneumonia with interstitial lung disease, radiation pneumonia, and immune-related pneumonia during the screening period, Presence of active tuberculosis, pneumoconiosis or grade 2 other type of pneumonia, or pulmonary function tests confirming severely impaired pulmonary function;
* Severe bone damage due to tumor bone metastasis may occur at present or after randomization;
* Active or uncontrolled serious infection (≥grade 2 infection of common toxicity criteria for adverse events (CTC AE)) or fever of unknown origin > 38.5°C;
* The third space effusion (including pleural effusion, abdominal effusion or pericardial effusion), poor clinical control or the need for local symptomatic treatment such as puncture and drainage;
* Known impaired gastrointestinal (GI) function or known GI diseases that may significantly affect the absorption or metabolism of oral drugs.

Previous history of major surgery in the digestive tract (esophagus, gastrointestinal tract) that may alter the absorption or inability to swallow drugs in the study treatment;

* Toxicity of previous antitumor therapy, except alopecia, pigmentation, clinically insignificant laboratory abnormalities) has not recovered to grade 1, and peripheral nerve toxicity has not recovered to grade 2 ( CTCAE v5.0);
* Human immunodeficiency virus (HIV) antibody positive, liver cirrhosis or active viral hepatitis;
* Active syphilis;
* Patients with renal failure requiring hemodialysis or peritoneal dialysis;
* Poor diabetes control [fasting blood glucose (FBG)> 10 mmol/L];
* Previous history of organ transplantation or readiness to undergo organ transplantation;
* Weight of <40 kg and BMI of <18.5 kg/m2, or weight loss of> 5% within 3 months before enrollment;
* Major surgical treatment or significant traumatic injury within 4 weeks prior to the first dose of this study;
* Receiving palliative radiotherapy with local lesions within 2 weeks before the first dose of this study;
* Pregnant or lactating subjects;
* With the combination of other primary malignancies
* Serious mental or mental illness or history of substance abuse or serious alcohol abuse;
* Known allergy to the investigational medicinal product or any ingredient in the formulation;
* Any other significant clinical abnormality or disease that the investigator considers poses a risk to subject safety or interferes with the medication and evaluation of the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Baseline up to 3 years
  Time from subject randomization (first treatment) to first disease progression or death from any cause, whichever occurred first, was assessed by an independent Review Committee (IRC) per Response evaluation criteria in solid tumors (RECIST) 1.1.

SECONDARY OUTCOMES:
Overall survival (OS) | Baseline up to 3 years
  From randomization to the time of death from any cause.
Objective mitigation rate (ORR) | Baseline up to 3 years
  According to RECIST 1.1 criteria, proportion of patients with confirmed tumor volume reduction to pre-specified values and maintained minimum requirements
  , namely the proportion of patients with complete response (CR) and partial response (PR).
Duration of Response (DOR) | Baseline up to 3 years
  From the time of tumor first evaluated as complete or partial response to the time of first disease progression or death from various causes.
Disease control rate (DCR) | Baseline up to 3 years
  According to RECIST 1.1 criteria, proportion of patients with confirmed tumor volume reduction to pre-specified values and maintained minimum requirements
  , namely the proportion of patients with CR, PR and stable disease (SD).
Time to response (TTR) | Baseline up to 3 years
  Time from patient randomization (first treatment) to first response per RECIST 1.1 criteria
Patient-reported outcome (PRO) | Baseline up to 3 years
  Reports of their health status directly from patients
Abnormal laboratory test indicators | From the subject signed the informed consent form to 30 days after the last dose
  The occurrence of laboratory test indicators exceed the normal range
Adverse event rate | From the subject signed the informed consent form to 30 days after the last dose
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs)
Time to Maximum Plasma Concentration (Tmax) | Pre-dose and 2 hours after D1553 administration on Day 1 of cycle 1 and cycle 3. Each cycle is 21 days.
  Time to maximum plasma concentration after dosing
Half life (t1/2) | Pre-dose and 2 hours after D1553 administration on Day 1 of cycle 1 and cycle 3. Each cycle is 21 days.
  Time required for plasma concentrations to drop by half

CONTACTS AND LOCATIONS:
Locations (85):
- China (85):
  - Anhui Province Hospital, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital,Capital Medical University, Beijing, Beijing Municipality
  - The Fifth medical center of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - The Southwest hospital of AMU, Chongqing, Chongqing Municipality
  - Army Medical Center, Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital Of Fujian Medical University, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - The Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - The Second Affiliated Hospital of Guilin Medical College, Guilin, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Yulin First People's Hospital, Yulin, Guangxi
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - The Second Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Hainan Provincial People's Hospital, Haikou, Hainan
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - The Affiliated Hospital of Chengde Medical College, Chengde, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tangshan People's Hospital, Tangshan, Hebei
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Jiamusi Tuberculosis Hospital(Jiamusi Cancer Hospital), Jiamusi, Heilongjiang
  - Anyang Tumor Hospital, Anyang, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Nanyang second general hospital, Nanyang, Henan
  - The First affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - The First Affiliated Hospital Of Xinxiang Medical Unerversity, Xinxiang, Henan
  - Xuchang Central Hospital, Xuchang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital Zhejiang University School of Medicine, Zhengzhou, Henan
  - Henan Provincial People's Hospita, Zhengzhou, Henan
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Zhongnan hospital of Wuhan University, Wuhan, Hubei
  - The Second Xiangya Hospital Of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The first people's hospital of Changzhou, Changzhou, Jiangsu
  - General Hospital of eastern theater command, Nanjing, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Jiangyin People's Hospital, Wuxi, Jiangsu
  - The Affiliated Hospital Of XuZhou Medical University, Xuzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shengjing hospital of China medical university, Shenyang, Liaoning
  - Shandong Cancer Hospitai, Jinan, Shandong
  - Jining First People's Hospital, Jining, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - The Second Affiliated Hospital of Shandong First Medical University, Tai’an, Shandong
  - Weifang people's Hospital, Weifang, Shandong
  - Weihai Municipal Hospital, Weihai, Shandong
  - Ruijin Hospital, Shanghai Jiaotong University School Of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Changzhi People's Hospital, Changzhi, Shanxi
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - The Second Affiliated Hospital of Air Force Medical University, Xian, Shanxi
  - The First Affiliated Hospital of Xi'An JiaoTong University, Xi’an, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The Affiliated Hospital Of Southwest Medical Unerversity, Luzhou, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - The second people's hospital of neijiang, Neijiang, Sichuan
  - Tianjin medical University cancer, Tianjin, Tianjin Municipality
  - The Affiliated Tumor Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang